CLINICAL TRIAL: NCT02329964
Title: Comparison of the Effectiveness of Rocuronium - Sugammadex With Succinylcholine-Cisatracurium-Neostigmine in Patients Undergoing Laser Microlaryngeal Surgery
Brief Title: Effectiveness of Sugammadex in LMS Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Seol Ju, Park, Resident, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LMS-sugammadex study KoreaUH
Record Dates: First submitted 2014-12-27; First posted 2015-01-01 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Relaxation
Keywords: Rocuronium; Sugammadex; Succinylcholine; Cisatracurium; Neostigmine; acceleromyography (TOF-Watch®)
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-S group (Experimental): Rocuronium-Sugammadex group
  1. Induction of anesthesia : 1% propofol 1.5-2.5 mg/kg with fentanyl 1.5 mcg/kg
  2. Muscle relaxant agent : Rocuronium 1mg/kg
  3. After endotracheal intubation : normal saline(0.025 ml/kg)
  4. Additive dose, for ensuring that neuromuscular blockade remains below T2 during surgery : Rocuronium 0.15mg/kg
  5. Relaxant agent reversal. at the the end of surgery : sugammadex 2mg/kg
  Interventions: Drug: Sugammadex
- S-C-N group (Active Comparator): Succinylcholine-Cisatracurium-Neostigmine group
  1. Induction of anesthesia :1% propofol 1.5-2.5 mg/kg with fentanyl 1.5 mcg/kg
  2. Muscle relaxant agent :Succinylcholine 1mg/kg
  3. After endotracheal intubation : Cisatracurium 0.08mg/kg
  4. Additive dose, for ensuring that neuromuscular blockade remains below T2 during surgery : Succinylcholine 10mg
  5. Relaxant agent reversal at the appearance of second TOF twitch (T2) : Neostigmine 0.2mg/kg with atropine 10 mcg/kg (for preventing side effects of neostigmine)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 2mg/kg was injected to patients to R-S group, as reversal of neuromuscular blockade.
  Other Names: Bridion
  Arms: R-S group
Drug: Neostigmine — Neostigmine (pyridostigmine) 0.2 mg/kg mg was injected to patients to S-C-N group, as reversal of neuromuscular blockade.
  Other Names: Pyridostigmine(Pyrinol)
  Arms: S-C-N group

SUMMARY:
This study is comparing of rocuronium-sugammadex and succinylcholine during LMS surgery that is characterized by short operation time, required intense paralysis and ambulatory setting, has not been investigated.

DETAILED DESCRIPTION:
Laser microlaryngeal surgery (LMS) requires brief and intense paralysis in the short operation time and the ambulatory setting.

The ideal muscle relaxant with rapid onset time, short duration of action and minimal side effects is not yet available.

Succinylcholine (SCC) is commonly used muscle relaxant for LMS because of its rapid onset time and short duration of action.

The use of SCC for tracheal intubation is usually followed by repeated small boluses or drip of SCC or small boluses of nondepolarizing muscle relaxants with intermediate duration.

As an alternative to SCC, the non-depolarizing neuromuscular blocking agent rocuronium can be used for LMS. The onset of rocuronium 1mg/kg is around 60s that is similar to SCC. However higher doses of rocuronium have a long duration of action; this is inappropriate in ambulatory surgery that requires rapid recovery of neuromuscular function and rapid turnover.

Sugammadex has recently been introduced as a selective relaxant-binding agent that allows for rapid reversal of rocuronium-induced neuromuscular blockade. Even profound neuromuscular block with rocuronium can be quickly antagonized with sugammadex.

After obtaining Institutional Review Board approval and written informed consent, 80 patients is enrolling in this study.

Patients is divided by two groups randomly as the Rocuronium-Sugammadex group(R-S group) and the Succinylcholine - Cisatracurium- Neostigmine group(S-C-N group) .

Anesthesia was induced with intravenous propofol 1.5-2.5 mg/kg, together with fentanyl1.5 mcg/kg After induction of anesthesia, neuromuscular monitoring is performed continuously at the adductor pollicis muscle with acceleromyography (TOF-Watch®).

Subsequently, in the R-S group, patients receive rocuronium 1mg/kg and in the S-C-N group, patients receive SCC 1mg/kg.

After T1 assessed as being zero by neuromuscular monitoring, endotracheal intubation is performed.

After endotracheal intubation, in the S-C-N group, cisatracurium 0.08mg/kg is injected and in the R-S group, the same volume of normal saline is injected.

Anesthesia is maintained with desflurane with air during the surgery. Additive dose of rocuronium 0.15mg/kg or SCC 10mg is given as necessary to ensure that neuromuscular blockade remains below T2 during surgery.

After the surgical procedure ends, patients receive sugammadex 2mg/kg in the R-S group, and pyridostigmine 0.2 mg/kg with atropine 10mcg/kg in the S-C-N group at the appearance of second TOF twitch (T2).

Patient will be assessed for the time to recovery of the TOF ratio to 0.9, surgical rating scale (1- extremely poor conditions, 2- poor conditions, 3- acceptable conditions, 4- good conditions, 5- optimal conditions), and anesthesia time.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist[ASA] class 1-3
* scheduled Laser microlaryngeal surgery under general anesthesia
* written informed consent

Exclusion Criteria:

* suspected difficult tracheal intubation
* disorder affecting neuromuscular blockade
* known or suspected significant renal dysfunction
* known or suspected severe hepatic dysfunction
* history of malignant hyperthermia
* allergy of opioids, neuromuscular blocking drugs or other medications used during general anesthesia
* contraindication to pyridostigmine and/or atropine
* pregnancy
* breast feeding
* body mass index > 27kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jangeun Cho, M.D.,Ph.D., Principal Investigator — Anesthesia and pain medicine department, Korea University Anam Hospital

REFERENCES:
- [Result] Lee C, Jahr JS, Candiotti KA, Warriner B, Zornow MH, Naguib M. Reversal of profound neuromuscular block by sugammadex administered three minutes after rocuronium: a comparison with spontaneous recovery from succinylcholine. Anesthesiology. 2009 May;110(5):1020-5. doi: 10.1097/ALN.0b013e31819dabb0. PMID 19387176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period : 2015.2.10 - 2015.6.30 Location : Korea University Medical Center Anam Hospital
Groups:
- R-S Group: Rocuronium-Sugammadex group
  1. Induction agent :
     * IV Propofol 1.5-2.5 mg/Kg and fentanyl 1.5mcg/kg
  2. During induction of anesthesia, as muscle relaxant agent
     * Rocuronium 1mg/kg
  3. After endotracheal intubation
     * normal saline(0.025 ml/kg)
  4. Additive dose, for ensuring that neuromuscular blockade remains below T2 during surgery
     * Rocuronium 0.15mg/kg
  5. Relaxant agent reversal. at the the end of surgery.
     * sugammadex 2mg/kg
- S-C-N Group: Succinylcholine-Cisatracurium-Neostigmine group
  1. Induction agent :
     * IV Propofol 1.5-2.5 mg/Kg and fentanyl 1.5mcg/kg
  2. During induction of anesthesia, as muscle relaxant agent
     * Succinylcholine 1mg/kg
  3. After endotracheal intubation,
     * Cisatracurium 0.08mg/kg
  4. Additive dose, for ensuring that neuromuscular blockade remains below T2 during surgery
     * Succinylcholine 10mg
  5. Relaxant agent reversal. at the appearance of second TOF twitch (T2).
     * Neostigmine 0.2 mg/kg with atropine 10μg/kg (for preventing side effects of neostigmine)
Period: Overall Study
Arm/Group | R-S Group | S-C-N Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R-S Group | S-C-N Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 32 | 69
  >=65 years | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 52 (15) | 50 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Recovery of T1 to 90%
Description: we measure the time from the end of surgery to recovery of the TOF 0.9. The end of surgery is defined as the time when the direct laryngoscope, aided by an operation microscope, is removed.
Time Frame: from the end of surgery(when the surgeon removes the suspension laryngoscope ) to time when the TOF ratio is 0.9, up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
seconds | 377 [334 to 435] | 240 [180 to 360]

2. Primary Outcome: Surgical Rating Score
Description: describe by surgeon under his subjective opinion.
  1 - extremely poor conditions 2- poor conditions 3- acceptable conditions 4- good conditions 5- optimal conditions
Time Frame: during surgery
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
score | 5.0 [5.0 to 5.0] | 5.0 [4.0 to 5.0]

3. Primary Outcome: Addition of Neuromuscular Blocking Agents
Description: Repeated small boluses or drip of Succinylcholine, or small boluses of nondepolarizing muscle relaxants with intermediate duration are usually followed.
  In this protocol, cisatracurium was injected after intubation to maintain neuromuscular blockade during surgery.
  We measure the requirement of additive dose of neuromuscular blocker to ensure that neuromuscular blockade remains below T2 during surgery
Time Frame: during surgery
Measure: Number; unit: participants
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
participants | 0 | 20

4. Secondary Outcome: Time to Extubation
Description: We expected the emergence time is shorter in R-S group than S-C-N group. So we measure the time from the end of surgery to recovery of the TOF 0.9, and the time from the end of surgery to extubation
Time Frame: from the end of surgery to extubate a tracheal tube
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
seconds | 430 [366 to 510] | 380 [286 to 495]

5. Other Pre Specified Outcome: Length of Stay in te Operating Room
Description: LMS surgery has short operation time and ambulatory setting. So the length of stay in the operating room will have significant. We expected the lengh of stay in the operating room is more shorter in R-S group than S-C-N group.
Time Frame: time from in to out of the operating room
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
minutes | 31.0 (7.7) | 38.6 (7.5)

6. Other Pre Specified Outcome: Anesthesia Time
Description: time from propofol injection to extubation
Time Frame: from the anesthesia start to end
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
minutes | 28.4 (7.5) | 35.2 (7.0)

7. Primary Outcome: Recovery of T1 to 10%
Description: we measure the time from the end of surgery to recovery of the TOF 0.1. The end of surgery is defined as the time when the direct laryngoscope, aided by an operation microscope, is removed.
Time Frame: from the end of surgery to time when the TOF ratio is 0.1, up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
seconds | 271 [183 to 330] | 190 [105 to 300]

8. Secondary Outcome: Time to First Spontaneous Breath
Description: time from end of surgery to first spontaneous breaths
Time Frame: from end of surgery to first spontaneous breaths
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
seconds | 263 [175 to 334] | 240 [70 to 325]

9. Secondary Outcome: Time to Eye Opening
Description: We expected the emergence time is shorter in R-S group than S-C-N group. So we measure the time from the end of surgery to opening of the eyes to verbal commands.
Time Frame: from end of surgery to opening of the eyes to verbal commands
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | R-S Group | S-C-N Group
Number analyzed (Participants) | 40 | 40
seconds | 340 [200 to 517] | 300 [180 to 420]

ADVERSE EVENTS:
Arm/Group | R-S Group | S-C-N Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The surgical rating score was assessed on the basis of the degree of laryngx exposure. This was influenced not only by neuromuscular relaxation but also by anatomical factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No